CLINICAL TRIAL: NCT01017367
Title: Phase 2, Multi-dose, Double-blind, Placebo-controlled, Randomized, Multicenter Study of MDX-1100 (Anti-CXCL10 Human Monoclonal Antibody) in Combination With Methotrexate in Subjects With Active Rheumatoid Arthritis (RA)
Brief Title: Study of MDX-1100 (Anti-CXCL10 Human Monoclonal Antibody) in Combination With Methotrexate in Subjects With Active Rheumatoid Arthritis (RA)
Acronym: MDX1100-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDX1100-04; IM129-003 (Other: BMS)
Record Dates: First submitted 2009-11-16; First posted 2009-11-20 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; inflammatory joint disease
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — MDX-1100

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MDX-1100 (Experimental): MDX-1100 10 mg/kg administered i.v. over 60 minutes on days 1, 15, 29, 43, 57, and 71
  Interventions: Drug: MDX-1100
- Placebo (Placebo Comparator): Placebo (saline) administered i.v. over 60 minutes on days 1, 15, 29, 43, 57, and 71
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDX-1100 — MDX-1100 10 mg/kg i.v. over 60 minutes on days 1, 15, 29, 43, 57 and 71
  Other Names: Anti CXCR4 Monocolonal anti-body, anti-IP-10
  Arms: MDX-1100
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to:

1. determine the American College of Rheumatology (ACR) 20 response rate at Day 85 in subjects with active rheumatoid arthritis(RA) administered MDX 1100 with methotrexate (MTX); and
2. determine the tolerability and safety of multiple doses of MDX-1100 in combination with MTX in subjects with active RA.

DETAILED DESCRIPTION:
This Phase 2, double-blind, placebo-controlled, randomized, multi-dose, multicenter study of MDX 1100 (anti CXCL10 human monoclonal antibody) in combination with MTX in subjects with active RA. All subjects will continue to receive stable doses of MTX (10 to 25 mg weekly) during the study. Eligible subjects (n=70) will be randomized to receive either placebo (n=35) or MDX-1100 (n=35) at 10 mg/kg intravenously, every other week for a total of 6 doses. Concomitant treatment with stable doses of prednisolone (≤ 10 mg/d, or equivalent) and non-steroidal anti-inflammatory drugs (NSAIDS) and analgesic drugs will be permitted during the study, however, the dose should not be changed until after the Day 85 assessment has been completed unless rescue therapy is required for significant worsening symptoms prior to Day 85. After Day 85, subjects will be followed until Day 141 only for safety and pharmacokinetics, and changes to baseline medications or addition of new medication will be permitted at the Investigator's discretion. Non-steroid anti-inflammatory drugs (NSAIDS) or analgesics should not be administered prior to disease activity assessments on study visit days.

Subjects withdrawn prior to Day 85 will be followed for safety for 70 days following their last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the ACR criteria for RA
* Must have active RA, characterized by at least 6 out of 66 swollen joints and 6 out of 68 tender joints, and at least 2 of the following: a serum C-reactive protein level greater than the upper limit of normal, an erythrocyte sedimentation rate >= 28 mm per hour, or morning stiffness > 45 minutes
* Seropositive for rheumatoid factor, as defined by a plasma rheumatoid factor level of at least 20 IU per milliliter and/or be seropositive for anti-cyclic citrullinated peptide antibody
* Must be on MTX (10 to 25 mg weekly) for at least 6 months receiving a stable dose for 42 days before randomization and no anticipated change in MTX dose while on study

  * Low-dose corticosteroids and NSAIDs are permitted at study entry and must have been stable for at least 28 days before randomization
  * All other disease modifying non-biologic anti-rheumatic drugs (DMARDs) must have been discontinued at least 28 days prior to randomization except for leflunomide (discontinued at least 60 days before randomization). Etanercept (discontinued at least 28 days prior to randomization) and infliximab, adalimumab, and abatacept (discontinued at least 56 days prior to randomization)
* Screening laboratory values

  * Hemoglobin ≥ 8.5 g/dL
  * White blood cell (WBC) ≥ 3000/mm³
  * Neutrophils ≥ 1.5x10(9)/L
  * Platelets ≥ 125x10(9)/L
  * Serum creatinine < 2 mg/dL
  * Aspartate aminotransferase (AST) ≤ 2xULN
  * Alanine aminotransferase (ALT) ≤ 2xULN
* Women must be postmenopausal (> 12 months without menses) or surgically sterile or using effective contraception for at least 4 weeks prior to the anticipated Visit 2 date and agree to continue contraception for the duration of their participation in the study
* Sexually active male subjects must use a barrier method of contraception during the course of the study.

Exclusion Criteria:

* Prior treatment with B cell depleting therapy
* Any other monoclonal antibody or immunoglobulin-based fusion proteins ≤ 8 weeks prior to randomization
* Any other experimental treatment ≤ 4 weeks prior to randomization
* Primary or secondary immunodeficiency
* Any other autoimmune disease other than RA (except concurrent Sjogren's syndrome or hypothyroidism)
* Complications of RA including:

  * Active rheumatoid vasculitis
  * Bed bound or wheelchair bound
  * Clinically significant pulmonary fibrosis
  * Felty's syndrome
* Any history of malignancy, excluding adequately treated and cured basal or squamous cell carcinoma of the skin, or cervical carcinoma in situ
* Active major psychiatric disease
* Evidence of acute or chronic infection
* Clinically significant cardiac disease requiring medication, unstable angina, myocardial infarction within 6 months of randomization, or congestive heart failure
* Arrhythmia requiring active therapy, with the exception of clinically insignificant extrasystoles, or minor conduction abnormalities;
* History of cerebrovascular disease requiring medication/treatment;
* Concomitant anticoagulation therapy or a known bleeding disorder
* Seizure disorder requiring active therapy
* Known drug or alcohol abuse
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
ACR 20 Response rate | 85 days

SECONDARY OUTCOMES:
Safety and tolerability will be monitored by physical exam, laboratory tests, electrocardiograms, chest x-ray and adverse events experienced and reported by the patient | 141 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- Romania (9):
  - Brasov Clinical County Emergency Hospital Rheumatology Department, Brasov
  - "Dr. Carol Davila" Central Military Emergency Clinical Hospital, Bucharest
  - Sana Medical Center, Bucharest
  - "Sf. Maria" Clinical Hospital, Department of Internal Medicine and Rheumatology, Bucharest
  - "Sf. Pantelimon" Emergency Clinical Hospital, Bucharest
  - Cluj Emergency County Clinical Hospital Rheumatology Department, Cluj-Napoca
  - Rehabilitation Hospital, Rheumatology Department, Iași
  - Targu-Mures County Clinical Hospital Rheumatology Department, Târgu Mureş
  - SC Excentric Company SRL, Rheumatology Department, Timișoara
- Ukraine (9):
  - M. Gorky National Medical University, Donetsk
  - V.K. Gusak Institute of Urgent & Reconstructive Surgery within the Academy of Medical Sciences of Ukraine, Hospital Therapy and Rehabilitation Clinic, Donetsk
  - Kharkiv Medical Academy of Postgraduate Education, Department of Cardiology and Functional Diagnostics, Clinical Facility: City Clinical Hospital #8, Kharkiv
  - Kyiv City Oleksandrivska Clinical Hospital, Rheumatology Department #2, Kyiv
  - O.O. Bogomolets National Medical University, Department of Internal Diseases Propedeutics #2, Clinical facility: City Clinical Hospital #3, Kyiv
  - Danylo Halytsky Lviv National Medical University, Department of Clinical Immunology and Allergology, Clinical Facility: Lviv Regional Clinical Hospital, Rheumatology Department, Lviv
  - Danylo Halytsky Lviv National Medical University, Department of Internal Diseases #2, Dermatology and Venerology within the Faculty of Continuing Education, Clinical facility: City Clinical Hospital #4, Rheumatology Department, Lviv
  - Public Institution O.I. Minakov City Clinical Hospital #9, Rheumatology Department, Odesa
  - Zaporizhya State Medical University, Department of Internal Diseases #2, Clinical facility: Medical and Sanitary Unit within the State-Owned Company "Radioprylad", Zaporizhya

REFERENCES:
- [Derived] Yellin M, Paliienko I, Balanescu A, Ter-Vartanian S, Tseluyko V, Xu LA, Tao X, Cardarelli PM, Leblanc H, Nichol G, Ancuta C, Chirieac R, Luo A. A phase II, randomized, double-blind, placebo-controlled study evaluating the efficacy and safety of MDX-1100, a fully human anti-CXCL10 monoclonal antibody, in combination with methotrexate in patients with rheumatoid arthritis. Arthritis Rheum. 2012 Jun;64(6):1730-9. doi: 10.1002/art.34330. Epub 2011 Dec 6. PMID 22147649